CLINICAL TRIAL: NCT00005402
Title: Transfusion Associated HCV in a Pediatric Population
Status: Completed | Type: Observational
Sponsor: Naomi Luban (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Naomi Luban, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 4319; R01HL056060 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2002-04

CONDITIONS: Transfusion-induced HCV and HGV Infection

SUMMARY:
To identify a large cohort of children transfused in the decade prior to second-generation anti-hepatitis C virus (HCV) donor screening (1982-1992). This will not only identify cases for the study of persistent infection and chronic hepatitis in children, but will allow for the determination of the annualized risk of transfusion-associated hepatitis (TAH) infection in children, data that are not currently available.

DETAILED DESCRIPTION:
BACKGROUND:

Accumulating data indicate that 70 to 80 percent of adults infected with the hepatitis C virus (HCV) develop persistent infection that may be associated with chronic hepatitis, cirrhosis, hepatocellular carcinoma and end-stage liver disease. Despite these potential mortal outcomes, the progression is indolent, and serious chronic sequelae may not occur for 10 to 50 years, by which time many transfused adults have died of unrelated causes. Infants and children, on the other hand, are far more likely to survive their transfusion episode, to have a long life span after HCV acquisition and, by inference, to experience the decades-long evolution to HCV-related cirrhosis and hepatocellular carcinoma.

DESIGN NARRATIVE:

The years 1982-1992 have been selected because TAH incidence in adults was still high at that time and because all subjects would be under age 15 at enrollment and unlikely to have been exposed to sexual contact or IV drug use. Maternal testing is performed to exclude perinatal transmission. Sixty-five hundred children who meet the eligibility criteria of the study have been transfused at Children's National Medical Center (CNMC) during this period, and archival serum specimens are available for 22 percent. The total eligible cohort is contacted and asked to provide a blood sample that is tested for antibodies to HCV and to the newly discovered hepatitis G virus (HGV). Subjects found antibody positive on initial screen are enrolled in long-term followup that includes serial determinations for alanine aminotransferase (ALT), other liver-related assays, viral serology with confirmatory testing, PCR for HCV and HGV RNA, HCV genotyping and, in those with evidence of chronic hepatitis, liver biopsy. Biopsy may also be performed on a subset with chronic viremia, but normal ALT, pending approval of an advisory panel of liver experts. A serum repository will be established for evaluation of new diagnostic methods for HCV, HGV, and other etiologic agents of posttransfusion hepatitis.

This study will determine the minimal rate of transfusion-induced HCV and HGV infection and will allow for an annualized incidence estimate and a determination of the national burden of transfusion-induced hepatitis virus infection in children, a value that is currently unknown. In addition, by use of archival samples and the interval from transfusion to testing, the study will determine the duration of infection and rate of viral persistence. Finally, prospective followup with liver biopsy will establish the extent of disease in those chronically infected. If persistent infection and chronic liver disease are as common in children as in adults, this would have major implications for anti-viral therapy programs and might shift treatment emphasis to pediatric populations where response rates might be higher and where long-term benefit would be greater.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-05; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)